CLINICAL TRIAL: NCT00348972
Title: Assessment of Safety and Tolerability of Lantus® (Insulin Glargine) in Subjects With Impaired Fasting Glucose (IFG) or Impaired Glucose Tolerance (IGT)
Brief Title: Lantus in Prediabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOE901/1021; HOE901
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2006-07-06 (Estimated); Status verified 2006-07

CONDITIONS: Hyperglycemia; Diabetes Mellitus
Keywords: Glargine; prediabetes; impaired glucose tolerance; impaired fasting glucose
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Prediabetic State; Glucose Intolerance | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Lantus® (insulin glargine)

SUMMARY:
To assess the safety, tolerability, and efficacy of Lantus® (insulin glargine) in prediabetes (IFG or IGT).

ELIGIBILITY:
Inclusion Criteria:

* Hyperglycemia (either IGT , IFG, or untreated type 2 diabetes)
* HbA1c < 7.0%
* BMI < 40kg/m2
* Able to perform moderate stationary bicycle exercise

Exclusion Criteria:

* Chronic pharmacologic treatment for hyperglycemia, past or present
* CAD
* serum creatinine > 2.0mg/dL
* BP > 180/105
* History of hypoglycemia unawareness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-02

PRIMARY OUTCOMES:
Efficacy: 8-point blood glucose measurements.
Safety / tolerability: hypoglycemia

SECONDARY OUTCOMES:
Blood glucose in response to exercise.
Fasting supine levels of counterregulatory hormones

CONTACTS AND LOCATIONS:
Overall Officials: Peter JOHNSTON, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com